CLINICAL TRIAL: NCT02948608
Title: Effectiveness and Patient-reported Outcomes in Patients With Spondyloarthropathies Treated With Biological Agents
Brief Title: Clinical Characteristics of Importance to Outcome in Patients With Spondyloarthritis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Svendborg Hospital (Other)
Collaborators: Odense University Hospital (Other); Parker Research Institute (Other); Spine Centre of Southern Denmark (Other)
Responsible Party: Principal Investigator, Rikke Asmussen Andreasen, MD, Svendborg Hospital
Other Study IDs: S-20160094; R-144-A4136 (Other Grant/Funding Number: The Danish Rheumatism Association)
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Spondyloarthropathy
Keywords: spondyloarthropathy; ankylosing spondylitis; spinal diseases; spondylitis; spondylarthritis; psoriasis; uveitis; joint diseases
MeSH Terms: conditions — Spondylarthropathies; Spondylitis, Ankylosing; Spinal Diseases; Spondylitis; Spondylarthritis; Psoriasis; Uveitis; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A Biobank will be established in connection with the routine blood samples taken at baseline (~ 90 ml). The blood samples will be handled and registered by research laboratory technicians at the laboratory department, and stored at Odense University Hospital, Denmark (in the cold store)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of the study is to investigate extra-articular manifestations, pain mechanisms, patient-reported outcomes, comorbidities and association between these conditions in patients with spondyloarthropathy (SpA) treated with Biologics. Further, to assess the predictive value of baseline pain profile on treatment outcome after ≥ 3 months.

DETAILED DESCRIPTION:
Patients with spondyloarthropaty, who initiate or switch biologics in routine care due to an active disease state, will be enrolled in this observational study.

The overall aim is to investigate extra-articular manifestations, pain mechanisms and patient-reported outcomes and elucidate if these factors - independently or by interaction - influence treatment response after ≥ 3 months. Patients will have a baseline visit, an eye examination and a follow up visit after ≥ 3 months. Clinical examinations will be performed at both time points and include:

1. Clinical examination (the spinal movement)
2. Assessment of pain mechanisms by clinical evaluation (BASDAI, tender points,) and pain questionnaires (PainDETECT).
3. The SPARCC Enthesitis Index will be used to enthesitis count.
4. Interview and questionnaires regarding lifestyle, comorbidity, function and quality of life
5. Blood samples
6. Urine samples
7. Stool samples

Clinical as well as patient-reported and observer-based outcomes will be described for the overall study population and the prognostic influence of extra-articular manifestations, comorbidity and pain mechanisms will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with SpA
* ≥18 years of age at time of consent
* Ability and willingness to give written informed consent and to meet the requirements of this protocol
* Patients must have a history of active disease and a BASDAI >40 (10-100) or elevated C-reactive protein, despite current or previous NSAIDs therapy

Exclusion Criteria:

* Age < 18 years
* No consent
* Pregnancy
* Active or latent TB
* Diagnosed Human immunodeficiency virus
* Diagnosed hepatitis
* Current or past malignant disease
* Recurrent or chronic infection (viral, fungal or bacterial)
* Multiple sclerosis
* Heart failure (NYHA class III/IV)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ≥ 18 years and diagnosed with any disease of the SpA spectrum, and about to initiate or switch biological treatment. We use the Assessment of Spondyloarthritis International Society (ASAS) criteria for SpA, and the Modified New York criteria for ankylosing spondylitis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Ankylosing Spondylitis Disease Activity Index BASDAI 50 % | ≥ 3 month from baseline
  composite measures of improvement in disease state (50% improvement)

SECONDARY OUTCOMES:
Change in Ankylosing Spondylitis Disease Activity Score (ASDAS) | ≥ 3 month from baseline
  composite measures of improvement in disease state

OTHER OUTCOMES:
To analyse the influence of PDQ score on the treatment response | ≥ 3 month from baseline
  we analyse if the painDETECT questionnaire score (PDQ) at baseline can influence on treatment outcome
Characterisation of the extra-articular manifestations in SpA patients | at baseline and ≥ 3 months from baseline
  To characterise the extra-articular manifestations according to ASAS criteria
Change in Bath Akylosing Spondylitis Functional Index (BASFI) | ≥ 3 month from timeline
Change in Spondylitis Consortium of Canada enthesitis score (SPARCC) | ≥ 3 month from baseline
Change in score of Medical Outcomes Study Questionnaire (SF-36) for mental and physical Health | ≥ 3 month from baseline
Change in plasma calprotectin (microg/L) | ≥ 3 month from baseline
Change in the Simple Clinical Colitis Activity Index (SCCAI) | ≥ 3 month from baseline
  composite measures of improvement in disease state
Change in the Harvey Bradshaws Activity Index (HBAI) | ≥ 3 month from baseline
  composite measures of improvement in disease state (Crohns disease)
Change in fecal calprotectin (mg/kg) | ≥ 3 month from baseline
Change in C-Reactive Protein, CRP (mg/L) | ≥ 3 month from baseline
Change in Visual Analogue Scale (VAS) (0-100 mm) of fatigue | ≥ 3 month from baseline
Change in Visual Analogue Scale (VAS) (0-100 mm) of fatigue of pain | ≥ 3 month from baseline
Change in Visual Analogue Scale (VAS) (0-100 mm) of global disease impact | ≥ 3 month from baseline
Withdrawal of treatment due to adverse event during the study period | ≥ 3 month from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Inger Marie J Hansen, MD, DmSci, Study Chair — Svendborg Hospital
Locations (1):
- Odense University Hospital, Svendborg Hospital, Svendborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andreasen RA, Kristensen LE, Ellingsen T, Christensen R, Baraliakos X, Wied J, Aalykke C, Ulstrup T, Schiottz-Christensen B, Horn HC, Emamifar A, Duerlund B, Fischer L, Hansen IMJ. Clinical characteristics of importance to outcome in patients with axial spondyloarthritis: protocol for a prospective descriptive and exploratory cohort study. BMJ Open. 2017 Jul 10;7(7):e015536. doi: 10.1136/bmjopen-2016-015536. PMID 28698330